CLINICAL TRIAL: NCT02149888
Title: A Pilot Study of Daily TDF/FTC-based PrEP Among High-risk Toronto MSM:The PREPARATORY-5 Study
Brief Title: PRe-Exposure Prophylaxis Acceptability & Readiness Assessments for Toronto gaY, Bisexual and Other Men Who Have Sex With Men-5
Acronym: PREP-5
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Hassle Free Clinic (Unknown); Maple Leaf Research (Other); Toronto Metropolitan University (Other); AIDS Committee of Toronto (Other); Canadian AIDS Treatment Information Exchange (Unknown); Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PREPARATORY-5
Record Dates: First submitted 2014-05-12; First posted 2014-05-29 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: HIV; Human Immunodeficiency Virus
Keywords: HIV; Pre-Exposure Prophylaxis; PrEP; Human Immunodeficiency Virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Tenofovir; Emtricitabine; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tenofovir/emtricitabine (Experimental): MSM receiving once daily TDF/FTC-based (Truvada®) pre-exposure prophylaxis
  Interventions: Drug: Tenofovir/emtricitabine

INTERVENTIONS:
Drug: Tenofovir/emtricitabine — Once daily Tenofovir/emtricitabine (Truvada®)
  Other Names: Truvada®

SUMMARY:
Canada continues to see an unrelenting stream of new HIV diagnoses, with a disproportionate burden among gay, bisexual, and other MSM in major centers such as Toronto. Pre-exposure prophylaxis (PrEP) with oral, daily tenofovir/emtricitabine (TDF/FTC, Truvada®) is a novel biomedical approach to HIV prevention shown in the iPrEx trial to be safe and efficacious in reducing HIV acquisition by 44% among MSM, when provided in a comprehensive package of HIV prevention interventions including counseling, testing/treatment of sexually transmitted infections (STIs), and condoms. There is now widespread mobilization to assess the feasibility of PrEP roll-out worldwide, with urgent calls for 'demonstration projects' addressing real-world PrEP implementation issues.

PREPARATORY-5 is Canada's first PrEP demonstration project, and will examine real-world PrEP implementation issues including acceptability, effectiveness, impact on sexually transmitted infections, and strategies for supporting adherence outside the clinical trial setting. The investigators have also established a comprehensive community-based research program investigating the role of community-based organizations in PrEP implementation and delivery.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified man who has sex with men
* Age 18 years or older
* Able to communicate in both written and oral english
* HIRI-MSM score greater than or equal to 10
* At least one self-reported unprotected receptive anal sex act over the preceding 6 months
* Creatinine clearance greater than or equal to 60mL/min by Modified Diet in Renal Disease (MDRD) formula
* HIV un-infected at screening using standard ELISA and Western Blot testing

Exclusion Criteria:

* Clinical signs or symptoms suggestive of an HIV seroconversion illness within the last 3 months in the opinion of the investigator
* Use of pre- or post-exposure prophylaxis within the last 3 months
* Use of concomitant nephrotoxic drugs
* Use of concomitant immune modulatory drugs
* Hepatitis B surface antigen positivity
* Any condition or concomitant medication portending an increased risk of osteoporosis
* Enrollment in any other HIV prevention program or trial

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2014-10; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Participants' self-reported overall acceptability of PrEP | 12 months
  Participants' self-reported overall acceptability of PrEP over the full one-year follow-up period (including the use of the medication, clinic visits, and their impact on the participant's life) will be quantified using a Likert scale.
The level of community interest in PrEP | 12 months
  The level of community interest in PrEP will be measured by quantifying the volume, rate and HIV risk levels of patient referrals to the PrEP clinic from each key referral source

SECONDARY OUTCOMES:
Adherence to daily TDF/FTC-based PrEP | 12 months
  Adherence will be measured by self-report, pill count, and intra-RBC tenofovir diphosphate levels.
Time required by the patient, physician and research coordinator for each type of study visit. | 12 months
  The time required by the patient, physician and research coordinator will be measured for each type of study visit.
HIV infection | 12 months
  HIV infection will be detected using point-of-care tests, standard serology and HIV RNA testing.
Sexually transmitted infections | 12 months
  Testing will be performed at each study visit to screen for gonorrhea, chlamydia and syphilis infection, including pharyngeal swab cultures, rectal swab cultures and urine NAAT tests.
Burden of syndemic health problems | 12 months
  The burden of specific syndemic health problems (depression, social anxiety, substance abuse, sexual addiction, childhood sexual abuse, partner violence) will be quantified using standardized, validated psychometric tools.
Change in estimated glomerular filtration rate | 12 months
  Estimated by the Modified Diet in Renal Disease (MDRD) formula
Percentage change in bone mineral density at the lumbar spine and total hip | 12 months
Adverse events | 12 months
  Adverse events will be assessed at each visit via clinical assessment and laboratory monitoring (CBC, phosphate, urinalysis).
Pilot testing study instruments | 12 months
  Outcomes related to pilot testing study instruments will include numbers of minutes required and participant-reported acceptability for each procedure

CONTACTS AND LOCATIONS:
Overall Officials: Darrell Tan, MD FRCPC PhD, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Tan DHS, Schnubb A, Lawless J, Szadkowski L, Grennan T, Wilton J, Fowler S, Hart TA, Maxwell J, Raboud JM. Acceptability and tolerability of and adherence to HIV preexposure prophylaxis among Toronto gay and bisexual men: a pilot study. CMAJ Open. 2018 Dec 10;6(4):E611-E617. doi: 10.9778/cmajo.20180068. Print 2018 Oct-Dec. PMID 30530721
- [Derived] Wilton J, Noor SW, Schnubb A, Lawless J, Hart TA, Grennan T, Fowler S, Maxwell J, Tan DHS. High HIV risk and syndemic burden regardless of referral source among MSM screening for a PrEP demonstration project in Toronto, Canada. BMC Public Health. 2018 Feb 27;18(1):292. doi: 10.1186/s12889-018-5180-8. PMID 29486737